CLINICAL TRIAL: NCT00633971
Title: A Randomized Trial to Determine the Impact of Lymphedema Therapy on Quality of Life and Disease Severity in Patients With Post-Thrombotic Syndrome
Brief Title: Treatment Trial for Post-Thrombotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Chris Holmes, Associate Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRMS 08-065
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Post Thrombotic Syndrome
Keywords: Post thrombotic syndrome; Thrombosis; Deep vein thrombosis; Venous thrombosis; Edema; stasis ulcers
MeSH Terms: conditions — Postthrombotic Syndrome; Thrombosis; Venous Thrombosis; Edema; Varicose Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Complex lymphedema therapy (which includes compression stocking use)
  Interventions: Other: complex lymphedema therapy
- B (Other): Standard of care (compression stocking use at 30-40 mm Hg)
  Interventions: Other: complex lymphedema therapy

INTERVENTIONS:
Other: complex lymphedema therapy — Patients with established post thrombotic syndrome will be randomized to either compression stocking use or complex lymphedema therapy.

SUMMARY:
The purpose of this study is to determine if complex lymphedema therapy is effective in decreasing disease severity and improving quality of life in patients with post thrombotic syndrome.

DETAILED DESCRIPTION:
Post thrombotic syndrome (PTS) has a spectrum of disease manifestations ranging from minor skin discoloration to severe skin changes and venous ulcerations. Pain is often a prominent symptoms and PTS impairs patient quality of life. Prevention of PTS using compression stockings has been emphasized. There is a paucity of validated, effective treatments for PTS once the condition develops.

While the pathophysiology of PTS is incompletely understood, chronic venous hypertension and insufficiency may increase the workload of the lymphatic system and result in over-capacitance with secondary damage and eventual lymphatic insufficiency. In selected patients with PTS, we have noted a symptomatic improvement in patients who receive lymphedema therapy to the limb.

Complex lymphedema therapy (CLT) is a noninvasive treatment that includes four key components: meticulous skin care, manual lymph drainage, compression therapy, exercises and patient education for home management and continuation of the treatment. These techniques are designed to enhance lymph flow through intact cutaneous lymphatics and reduce swelling and restore function in the affected limb.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Diagnosis of post thrombotic syndrome.
* Median life expectancy of greater than 2 years.
* Previous history of lower extremity deep venous thrombosis.

Exclusion Criteria:

* Acute venous thrombosis of the lower extremity within the last 180 days.
* Unable to participate in lymphedema therapy due to monetary, physical or transportation limitations.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women and women in their first post-partum month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To determine if complex lymphedema therapy improves the quality of life in patients with post-thrombotic syndrome | 1 and 3 months
To determine if complex lymphedema therapy reduces disease severity in patients with post thrombotic syndrome | 1 and 3 months

SECONDARY OUTCOMES:
To assess side effects of lymphedema therapy when administered to patients with PTS | 1 and 3 months
To determine if selected biomarkers correlate with disease severity and response to lymphedema therapy in patients with post thrombotic syndrome | 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Chris E Holmes, MD, PhD, Principal Investigator — University of Vermont and Fletcher Allen Health Care
Locations (1):
- Fletcher Allen Health Care; Department of Hematology/Oncology, Burlington, Vermont, United States

REFERENCES:
- [Derived] Holmes CE, Bambace NM, Lewis P, Callas PW, Cushman M. Efficacy of a short course of complex lymphedema therapy or graduated compression stocking therapy in the treatment of post-thrombotic syndrome. Vasc Med. 2014 Feb;19(1):42-8. doi: 10.1177/1358863X14521883. PMID 24558028
- See also: Dedicated to improving the human condition affected by cancer, through research in the laboratory and in the clinic, cancer prevention and control research and programs, state-of-the art cancer diagnosis. — http://www.vermontcancer.org